CLINICAL TRIAL: NCT04762043
Title: EMG Voice Restoration
Brief Title: MyoVoice to Restore Natural, Hands-free Communication to Individuals With Vocal Impairments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Altec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EMG Voice Restoration
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-05

CONDITIONS: Rehabilitation of Speech and Language Disorders; Speech Disorders; Speech, Alaryngeal; Communication Aids for Disabled; Speech Perception; Speech Intelligibility
MeSH Terms: conditions — Language Disorders; Speech Disorders; Speech; Speech Intelligibility

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental and Reference Devices for Communication (Experimental): Each participant listens to speech produced by an experimental ("MyoVoice") and reference (electrolarynx) systems that are used to communicate. Participants rate the naturalness of the speech produced from each device (audio files presented in a randomized order). Duration: 30 mins to 1 hour.
  Interventions: Device: Experimental System: MyoVoice; Device: Reference System: Electrolarynx
- Development of Speech Corpora (No Intervention): Each participant produces a list of speech tasks that include syllables, phrases, reading passages, and open-ended questions using the MyoVoice system. Myovoice pitch and loudness recognition accuracy of speech is evaluated. Duration: 30 mins to 2 hours.

INTERVENTIONS:
Device: Experimental System: MyoVoice — Person-centric augmentative and alternative communication (AAC) system comprising a user-specific set of wearable sensors for capturing articulatory muscle activity and mobile software that provides real-time audible speech outputs.
  Arms: Experimental and Reference Devices for Communication
Device: Reference System: Electrolarynx — Hand-operated electromechanical device that operates as an artificial larynx to enable a person after laryngectomy to produce speech.
  Arms: Experimental and Reference Devices for Communication

SUMMARY:
This study will evaluate the ability of MyoVoice to replace natural speech. Referred to generally as an Augmentative and Alternative Communication (AAC) device, MyoVoice uses electrical signals recorded non-invasively from speech muscles (electromyographic, or EMG, signals) to restore communication for those with vocal impairments that resulted from surgical treatment of laryngeal and oropharyngeal cancers.

DETAILED DESCRIPTION:
Over 7.5 million people worldwide are unable to vocalize effectively. Among these individuals are cancer survivors who underwent oropharyngeal/laryngeal surgery and must rely on AAC systems such as text-to-speech applications or artificial voice prostheses as substitutes for their natural voice. Yet most of these devices struggle to convey the expressive attributes of speech (prosody), leading to poor comprehension and a lack of emotional content. The clinical trial will investigate the feasibility of MyoVoice-a novel AAC device that uses surface EMG signals to extract patterns for understanding vocabulary and expressive attributes from articulatory musculature during silently mouthed speech-to effectively restore conversational capabilities for individuals living with vocal impairments due to surgical treatment of laryngeal and oropharyngeal cancers. Patients who underwent a total laryngectomy will be asked to communicate with a conversational partner by silently mouthing words using MyoVoice. The device performance will be evaluated in terms of its ability to accurately and quickly translate articulatory muscle activity into audible speech. MyoVoice will also be compared to that of conventional electrolaryngeal speech aids (i.e., artificial larynx) to evaluate device ease-of-use, functional efficacy, and social reception.

ELIGIBILITY:
1. Individuals without Laryngectomy ("Controls")

   Inclusion Criteria:
   * Primary English speaker
   * No history of speech, language, cognitive, or hearing disorders
   * Normal hearing (able to pass a bilateral hearing screening using a threshold of 25 decibels (dB) hearing level (HL) at 125, 250, 500, 1000, 2000, 4000, and 8000 Hz based on the American Speech-Language-Hearing Association)
   * Capable of signed informed consent

   Exclusion Criteria:
   * Inability to understand spoken English or follow simple instructions
   * History of speech, language, cognitive, or hearing disorders
   * Inability to provide written informed consent
2. Individuals with Laryngectomy

Inclusion Criteria:

* At least 6 months S/P total laryngectomy
* Primary English speaker
* Proficient with an electrolarynx (EL)
* Sufficiently available and healthy to comply with multiple test sessions lasting 4-6 hours
* Capable of signed informed consent

Exclusion Criteria:

* Inability to understand spoken English or follow simple instructions
* Loss of adequate surface electromyographic (sEMG) sensor sites for recording from muscles of articulation due to cancer treatment
* Skin disorders or radiation/surgical scarring that prevent the use of medical-grade adhesive tapes for securing sensors
* Any other medical or psychological condition that is based on the opinion of investigations will prevent participation in the experiment (e.g., the candidate may have an illness that makes them fatigue easily or have difficulty to attend to visual cues)
* Inability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2023-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca DeLuca, Principal Investigator — Altec Inc.
Locations (1):
- Altec Inc., Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant demographics, summary data for all primary and secondary outcome measures, and study protocol will be made available.
Supporting Information: Study Protocol
Time Frame: Data will be made available within 6 months of study completion.
Access Criteria: Data access request will be made through conferencing.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Development of Speech Corpora | Experimental and Reference Devices for Communication
Started | 10 | 20
Completed | 10 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental and Reference Devices for Communication: Each participant listens to speech produced by an experimental ("MyoVoice") and reference (electrolarynx) systems that are used to communicate. Participants rate the naturalness of the speech produced from each device (audio files presented in a randomized order). Duration: 30 mins to 1 hour.
  Experimental System: MyoVoice: Person-centric AAC system comprising a user-specific set of wearable sensors for capturing articulatory muscle activity and mobile software that provides real-time audible speech outputs.
  Reference System: Electrolarynx: Hand-operated electromechanical device that operates as an artificial larynx to enable a person after laryngectomy to produce speech.
- Total: Total of all reporting groups
Arm/Group | Development of Speech Corpora | Experimental and Reference Devices for Communication | Total
Number analyzed (Participants) | 10 | 20 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 18 | 28
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (7.65) | 55 (7.30) | 42 (15.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 5 | 11 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 18 | 27
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 17 | 27
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 20 | 30

OUTCOME MEASURES:

1. Primary Outcome: Pitch Recognition Accuracy
Description: Percent accuracy between recognized (sEMG) and ground-truth (acoustic) estimates of fundamental frequency (perceptually known as vocal pitch). Accuracy is estimated on a continuous scale from 0 to 100%.
Time Frame: 30 mins to 2 hours
Population: The sEMG and acoustic data collected from participants in the "Development of Speech Corpora" arm were used to develop and evaluate an algorithm to predict vocal pitch (acoustic correlate: fundamental frequency) from sEMG data. Higher accuracy scores equate to better performance.
Measure: Mean (Standard Deviation); unit: Percent agreement to reference pitch
Arm/Group | Development of Speech Corpora | Experimental and Reference Devices for Communication
Number analyzed (Participants) | 10 | 0
Percent agreement to reference pitch | 7.70 (1.63) |

2. Primary Outcome: Loudness Recognition Accuracy
Description: Percent accuracy between recognized (sEMG) and ground-truth (acoustic) estimates of intensity level (perceptually related to vocal loudness). Accuracy is estimated on a continuous scale from 0 to 100%.
Time Frame: 30 mins to 2 hours
Population: The sEMG and acoustic data collected from participants in the "Development of Speech Corpora" arm were used to develop and evaluate an algorithm to predict vocal loudness (acoustic correlate: intensity) from sEMG data. Higher accuracy scores equate to better performance.
Measure: Mean (Standard Deviation); unit: Percent agreement to reference loudness
Arm/Group | Development of Speech Corpora | Experimental and Reference Devices for Communication
Number analyzed (Participants) | 10 | 0
Percent agreement to reference loudness | 12.1 (3.0) |

3. Primary Outcome: Speech Naturalness
Description: Percent naturalness between MyoVoice and electrolarynx speech samples. Speech naturalness is defined based on one's "preference for how [the audio] sounds in terms of rate, rhythm, intonation and voice quality." Naturalness is estimated on a continuous scale from 0 to 100%.
Time Frame: 30 mins to 1 hour
Population: Participants in the "Experimental and Reference Devices for Communication" rated the naturalness of each sample on a visual analog scale from 0 to 100, which 0 anchored at "least natural" and 100 anchored at "most natural." Higher naturalness scores equate to better performance.
Measure: Mean (Standard Deviation); unit: Percent of high naturalness ratings
Arm/Group | Development of Speech Corpora | Experimental and Reference Devices for Communication
Number analyzed (Participants) | 0 | 20
Percent of high naturalness ratings
  MyoVoice |  | 66.2 (22.6)
  Electrolarynx |  | 9.7 (19.8)
  Overall |  | 38.0 (35.4)
Statistical Analysis 1: Comparison: Experimental and Reference Devices for Communication; Test type: Superiority; p < .001, Mixed Models Analysis; Effect size used for mixed effects model is partial eta-squared (ηp2); Mean Difference (Final Values) = 56.55, 95% CI 2-sided [53.33 to 59.76], Standard Error of Mean 1.64

ADVERSE EVENTS:
Time Frame: 30 min - 2 hours
Arm/Group | Development of Speech Corpora | Experimental and Reference Devices for Communication
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/20
Other Adverse Events (participants affected / at risk) | 0/10 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/43/NCT04762043/Prot_001.pdf
  • Statistical Analysis Plan (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/43/NCT04762043/SAP_002.pdf
  • Informed Consent Form (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/43/NCT04762043/ICF_003.pdf